CLINICAL TRIAL: NCT01484522
Title: A Laboratory Study to Assess the Immunogenicity of Three Licensed Influenza A (H1N1) 2009 Monovalent Vaccines in HIV-1 Perinatally Infected Children and Youth
Brief Title: Laboratory Study of Licensed H1N1 Influenza Vaccines in HIV-1 Perinatally Infected Children and Youth
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1089; U01AI068632 (NIH)
Record Dates: First submitted 2011-09-29; First posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: HIV-1 Infection; H1N1; Influenza; Flu
Keywords: Influenza; Perinatal; immunogenicity; Monovalent vaccine; Children; Youth; H1N1; Adolescent; Flu
MeSH Terms: conditions — Influenza, Human | interventions — FluMist; Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group A: Influenza A 2009 Monovalent vaccine
  Interventions: Biological: FluMist
- Group B: Influenza A 2009 monovalent vaccine
  Interventions: Biological: Fluvirin
- Group C: Influenza A 2009 monovalent vaccine
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: FluMist — Administered at the manufacture's recommended dose
  Groups: Group A
Biological: Fluvirin — Vaccine administered at the manufacturer's recommended dose.
  Groups: Group B
Biological: Fluzone — Vaccine administered at manufacturer's recommended dose
  Groups: Group C

SUMMARY:
The purpose of this research study is to evaluate the immune response to the H1N1 influenza or "flu" vaccine. The "immune response" is how your body recognizes and defends itself against bacteria, viruses, and substances that may be harmful to the body.

HIV-1 infected children typically respond more poorly to vaccines compared to uninfected, healthy children and so this study hopes to learn whether or not the body will successfully produce enough antibodies (proteins that fight infection) that will prevent or fight the H1N1 flu virus. There is no information yet on the safety or immune response to this vaccine in children infected with HIV.

DETAILED DESCRIPTION:
HIV-infected children typically respond poorer to vaccines as compared to normal children. The FDA has currently approved several Influenza A 2009 monovalent vaccines to be used in children and adults. However, little data is available in perinatally infected youth. Therefore, knowledge of the immunogenicity of several of the licensed Influenza A 2009 monovalent vaccines in HIV-infected children and youth is critically important to address the health care needs of this vulnerable population. Efforts are currently underway to evaluate Influenza A 2009 monovalent vaccines in healthy children as well as other populations. This study will assess the immune response following receipt of three Influenza A monovalent vaccines in HIV-1 infected children and youth. Protection of HIV-1 infected children and youth from 2009 H1N1 Influenza A will require knowledge of immunogenicity of these new products in this population. The 2009 (H1N1) Influenza A virus is likely to infect a significant proportion of HIV-1 infected children and youth. Immunogenicity of licensed and commercially available Influenza A 2009 monovalent vaccines must be established in HIV-1 infected children in order to assure that this population is protected. Lack of a protective immune response would support the need for additional measures to protect this high risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Children and youth 6 months to <25 years of age at study entry.
2. HIV infection, defined as positive test results obtained from 2 different samples. Tests may include two of the same type OR two different types of tests listed below, as long as there are positive test results obtained from 2 different samples:

   * HIV-1 antibody (ELISA + WB), obtained at age >18 months
   * HIV-1 culture, any age
   * HIV-1 DNA PCR, any age
   * HIV-1 RNA PCR >10,000 copies/mL, any age
   * Neutralizable HIV-1 p24 antigen obtained >28 days of age
3. In the opinion of the investigator, the route of HIV-1 transmission is perinatally acquired.
4. Parent or legal guardian, youth of legal age, or subjects who are emancipated minors, who are willing and able to provide signed informed consent.
5. Planned receipt of one of the following FDA licensed Influenza A (H1N1) 2009 Monovalent Vaccines within 24 hours following study entry:

   * Group A: Influenza A (H1N1) 2009 Monovalent Vaccine (MedImmune FluMist®)
   * Group B: Influenza A (H1N1) 2009 Monovalent Vaccine (Novartis Fluvirin®)
   * Group C: Influenza A (H1N1) 2009 Monovalent Vaccine (Sanofi Pasteur Fluzone®) *OR has received one of the above vaccines within 4 hours prior to study entry.

Exclusion Criteria:

1. Has a history of probable or proven pandemic 2009 H1N1 Influenza A virus infection prior to study entry.
2. Has received seasonal FluMist vaccine within 2 weeks prior to study entry.
3. Has received any 2009 H1N1 vaccines prior to the day of entry.
4. Has received any immunoglobulin or blood products within 3 months prior to study entry.
5. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the study.
6. Use of anti-cancer chemotherapy or radiation therapy within the 36 months preceding study entry, or has immunosuppression as a result of an underlying illness or treatment (other than HIV-1 infection).
7. Has an active neoplastic disease.
8. Long term use of glucocorticoids, including oral or parenteral prednisone or equivalent (more than or equal to 2 mg/kg per day or more than or equal to 20 mg total dose) for more than 2 weeks in the past 6 months, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV-1 perinatally infected children and youth 6 months to 25 years of age.
  For inclusion into the study, if perinatal acquisition of HIV infection cannot be confirmed based on the child's medical record, it is acceptable to enroll the child if the investigator's assessment is that the most likely route of infection was perinatal.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The short term immune response following immunization with a licensed Influenza A (H1N1) 2009 Monovalent Vaccine administered as a single dose in perinatally HIV-1 infected children and youth aged >10 to <25 years. | 8 months
The short term immune response following second immunization with a licensed Influenza A (H1N1) 2009 Monovalent Vaccine in perinatally HIV-1 infected children > 6 months to < 10 years of age. | 8 months

SECONDARY OUTCOMES:
The immune response following first immunization with a licensed Influenza A (H1N1) 2009 monovalent vaccine in children aged > 6 months to < 10 years of age. | 8 months
Persistence of antibody responses 7 months after receipt of the first immunization with a licensed Influenza A (H1N1) 2009 monovalent vaccine. | 8 months
Immune responses with CD4+ cell count and timing of seasonal trivalent influenza vaccine (TIV). | 8 months
Immune responses with CD4 percent and timing of seasonal trivalent influenza vaccine (TIV). | 8 months
Immune responses with ARV use and timing of seasonal trivalent influenza vaccine (TIV). | 8 months
Immune responses with plasma HIV-1 RNA concentration and timing of seasonal trivalent influenza vaccine (TIV). | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Flynn, M.D., Study Chair — St. Jude Childrens Research Hospital
Locations (17):
- United States (16):
  - Univ. of Alabama Birmingham NICHD CRS (5096), Birmingham, Alabama
  - USC/Los Angeles County Medical Center NICHD CRS, Los Angeles, California
  - University of California San Francisco NICHD CRS (5091), San Francisco, California
  - University of Colorado Denver NICHD CRS (5052), Aurora, Colorado
  - University of Miami Pediatric/Perinatal HIV/AIDS (4201), Miami, Florida
  - University of South Florida Tampa (5018), Tampa, Florida
  - Chicago Children's CRS (4001), Chicago, Illinois
  - Children's Hospital of Boston NICHD CRS (5009), Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Wayne State University/Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - NJ Med School CRS (2802), Newark, New Jersey
  - New York University NY (5012), New York, New York
  - SUNY Stony Brook (5040), Stony Brook, New York
  - Jacobi Medical Center Bronx (5013), The Bronx, New York
  - The Children's Hospital of Philadelphia (6701), Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS (6501), Memphis, Tennessee
- University of Puerto Rico Pediatric HIV/AIDS Research (6601), San Juan, Puerto Rico